CLINICAL TRIAL: NCT00204932
Title: Effects of CLA Supplements on Body Weight and Fat Oxidation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004-0060
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Linoleic Acids, Conjugated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLA treatment (Active Comparator): The group randomized to Conjugated Linoleic Acid (CLA) treatment at 4 grams per day of 39% cis-9, trans-11 CLA; 39% trans-10, cis-12 CLA; and 22% safflower oil for 6 months
  Interventions: Drug: conjugated linoleic acid
- Placebo (Placebo Comparator): The group randomized to control received 4 g/d of safflower oil.
  Interventions: Drug: conjugated linoleic acid

INTERVENTIONS:
Drug: conjugated linoleic acid — 4 grams per day of 39% cis-9, trans-11 CLA; 39% trans-10, cis-12 CLA, and 22% safflower oil for 6 months

SUMMARY:
Conjugated linoleic acid (CLA) is form of fat found in dairy foods, beef and other natural sources. When given to small animals, decreases of body fat have been noted.. Although weight loss is the best treatment for overweight and obesity, it is difficult to maintain the loss in the long term. Because of this, treatment emphasis has turned to small weight losses obtained through non-restrictive diets and prevention of weight regain. This is a study to determine if 6 months of consumption a purified form of CLA will result in greater loss of body fat than control and to determine whether CLA consumption increases total fat oxidation, which would help explain why the weight loss occurs.

DETAILED DESCRIPTION:
Subjects were screened and then underwent baseline evaluation. The substudy evaluation measured 24-h energy expenditure and substrate utilization by using a whole-room indirect calorimeter. Dietary fat oxidation was measured by mixing [1-13C]oleate and D31-palmitate into a breakfast meal and then collecting breath carbon dioxide and urine to measure the end products of oxidation. Subjects were then provided either 4 g/d of 78% active CLA isomers (3.2 g/d: 39.2% cis-9,trans-11 and 38.5% trans-10,cis-12) or 4 g/d of safflower oil placebo as 1-g gel capsule supplements. The baseline evaluations were repeated 6 mo later.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-29.9 kg/m2
* Absence of a weight change of greater than 3 kg in the previous 6 months

Exclusion Criteria:

* Presence of a physical limitation to walking exercise
* Current or recent (6 months) enrollment in a commercial or self-prescribed weight loss program
* A history of metabolic disease-ie. renal, endocrine, hepatic or gastrointestinal disease that would impact the outcome of the study
* A history of a psychiatric or eating disorders Ÿ Presence of metal implants that would interfere with body composition analysis
* Fasting plasma cholesterol >300mg/dl or triglycerides above 500 mg/dl.
* Abnormal EKG

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2004-07; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dale A Schoeller, PhD, Study Chair — University of Wisconsin, Madison; Dale A Schoeller, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Result] Watras AC, Buchholz AC, Close RN, Zhang Z, Schoeller DA. The role of conjugated linoleic acid in reducing body fat and preventing holiday weight gain. Int J Obes (Lond). 2007 Mar;31(3):481-7. doi: 10.1038/sj.ijo.0803437. Epub 2006 Aug 22. PMID 16924272
- [Result] Close RN, Schoeller DA, Watras AC, Nora EH. Conjugated linoleic acid supplementation alters the 6-mo change in fat oxidation during sleep. Am J Clin Nutr. 2007 Sep;86(3):797-804. doi: 10.1093/ajcn/86.3.797. PMID 17823448

RESULTS

PARTICIPANT FLOW:
Groups:
- Conjugated Linoleic Acid: 4 grams per day of 78% CLA for 6 months
- Placebo: 4 grams per day of sunflower oil for 6 months
Period: Overall Study
Arm/Group | Conjugated Linoleic Acid | Placebo
Started | 24 | 24
Completed | 22 | 18
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Conjugated Linoleic Acid: 3 grams per day for 7 months
- Placebo: 3 grams per day of sunflower oil for 7 months
- Total: Total of all reporting groups
Arm/Group | Conjugated Linoleic Acid | Placebo | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (8) | 32 (7) | 33 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Fat Mass
Description: loss of fat mass, kg
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Conjugated Linoleic Acid | Placebo
Number analyzed (Participants) | 22 | 18
kg | -1.0 (2.2) | 0.7 (3.0)
Statistical Analysis 1: Comparison: Conjugated Linoleic Acid vs Placebo; Analysis of variance to test CLA not equal to placebo; Test type: Non-Inferiority or Equivalence — Power analysis was based on test-retest variance of body fat mass measure by DEXA; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: Conjugated Linoleic Acid vs Placebo; Pre- post treatment comparison o fat oxidation found that fat oxidation increased in CLA (4 +/- 8 g) and decreased in placebo (-7 +/- 11 g) groups during sleep. after 6 mo of supplementation; Test type: Superiority; p < 0.05, ANOVA

2. Secondary Outcome: Total Fat Oxidation
Description: 24 hour respiratory gas analysis
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Conjugated Linoleic Acid: 4 grams of 78% active CLA per day for 6 months
Arm/Group | Conjugated Linoleic Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 2/24 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conjugated Linoleic Acid (N=24) | Placebo (N=24)
blood chemistry: soluble vascular cell adhesion (Blood and lymphatic system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less